CLINICAL TRIAL: NCT05655546
Title: ImmunoCARE: Rapid, Accurate COVID Testing to Reduce Hospitalization of Immunocompromised Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: On May 13, 2024, the FDA released a communication that Cue Health tests should no longer be used.
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Cue Health (Unknown)
Responsible Party: Principal Investigator, Julia Moore Vogel, Program Director, Scripps Translational Science Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-22-8082
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Immunodeficiency; Immunosuppression; HIV Infections; Graft Versus Host Disease; Leukemia; Lymphoma; Cancer; Multiple Myeloma; Transplant; Age-Related Immunodeficiency
Keywords: COVID-19; Immunocompromised; Advanced Age; Medicare; Medicaid
MeSH Terms: conditions — Immunologic Deficiency Syndromes; HIV Infections; Graft vs Host Disease; Leukemia; Lymphoma; Neoplasms; Multiple Myeloma; COVID-19 | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Other): Participants in this group will complete the baseline study activities, as described above. Additionally, participants will be instructed to create a Cue Health account and download the Cue Health App. Using the app and the 10 Cue Health COVID-19 molecular tests that are provided (or Cue Health Flu+COVID molecular tests if available and FDA authorized), the participant will perform tests after exposure or if symptoms arise. Participants can also use the test for close contacts who are exposed to COVID-19 and/or have symptoms. If COVID-19 infection occurs, participants will have access to telemedicine to discuss further with a healthcare professional. When clinically indicated, medication for the treatment of COVID-19 (and/or Influenza in case of Cue Health Flu+COVID test availability) will be prescribed and delivered to the participants' delivery address. Participants can also seek care through other healthcare providers or not seek care, at their discretion.
  Interventions: Other: Access to Cue Health COVID-19 Remote testing and treatment for COVID-19
- Control Arm (No Intervention): Participants in the control group will complete the baseline study activities, as described above. If symptoms arise or COVID-19 infection occurs, participants will test and seek care as they normally would.

INTERVENTIONS:
Other: Access to Cue Health COVID-19 Remote testing and treatment for COVID-19 — Participants will receive at home COVID-19 test for themselves and others in their household.
  Arms: Intervention Arm

SUMMARY:
The investigators will examine whether a combination of at-home nucleic acid amplification tests, on-demand telemedicine, and delivery of prescriptions such as Paxlovid quickly after testing positive for COVID-19, can reduce severe outcomes and hospitalization of immunocompromised patients and those who are 65 years and older. They will also analyze whether these efforts lower the cost of care compared to standard of care.

DETAILED DESCRIPTION:
This study is a randomized control trial with 10,000 participants. Participation will last for a minimum of 3 months and maximum of 8 months, depending upon COVID-19 case rates. Half of participants will be randomized to the control group and continue their existing testing and healthcare practices. The remaining participants will be randomized into the intervention arm. Participants in the intervention will receive one Cue Cartridge Reader for the duration of the study and up to 10 Cue COVID Molecular tests per month for their own use and to share with others in their household. In the case that a Cue Flu+COVID Molecular Test is available through FDA EUA or other authorization, participants may be provided this multiplex test in lieu of the Cue COVID Molecular Test. All intervention participants will be asked to test themselves if they are exposed or when symptoms arise and share tests with members of their household who are exposed to COVID or symptoms arise. The primary outcome will be the number of hospitalizations. This study will also compare infection rates, ICU admissions, deaths, and cost of care between the control and intervention group. The hypothesis is that access to high sensitivity portable molecular testing and subsequent telemedicine and prescription delivery can significantly decrease hospitalization and thereby the cost of care.

Interested individuals will access the study via the MyDataHelps platform by web or app to complete the eligibility and informed consent process. Within the MyDataHelps experience, participants will complete study activities such as surveys and sharing of claims data. Participants who are randomized to the intervention group will have the option to use Cue Care should they test positive for COVID-19. Cue Care contracts licensed Healthcare providers to deliver telemedicine and treatment for COVID-19. In the case that the COVID Flu+COVID test is available, the intervention group will also have the option to use Cue Care should they test positive for Influenza.

To learn more and take the eligibility survey, visit https://ImmunoCARE.scripps.edu/

ELIGIBILITY:
Inclusion Criteria:

* Living in the United States
* 18 years or older
* Can read and understand English
* Use of smartphone with bluetooth, a camera and a compatible operating system (Android OS 9.0 or higher, Apple iOS 13.0 or higher)
* Vaccinated against COVID-19 (completed at least the initial course, e.g. at least 2 doses of -Moderna or Pfizer, one dose of J&J)
* Willing and able to participate in study interventions including:

  1. Use of smartphone, including camera and bluetooth
  2. Upload verification of diagnosis, if needed
  3. Completing Surveys
  4. Use of Cue Health App
  5. Use of MyDataHelps Web or App
* Immunocompromised due to disease or therapy, including:

  1. Symptomatic HIV
  2. Graft versus host disease
  3. Immunoglobulin deficiency/Immunodeficiency
  4. Immunosuppressive therapy
  5. Leukemia
  6. Lymphoma (Hodgkin or non-Hodgkin)
  7. Metastatic Cancer
  8. Multiple Myeloma
  9. Solid organ malignancy
  10. Transplant, hematopoietic stem cell
  11. Transplant, solid organ
* Age 1. 65 years and older

Option if under 65 to share claims data as a member of one of the following insurance providers:

1. Anthem BlueCross and BlueShield
2. Anthem BlueCross
3. Empire BlueCross BlueShield
4. Empire BlueCross
5. Wellpoint
6. Carelon
7. Unicare
8. Simply Healthcare Plans
9. National Government Services, Inc.
10. MMM
11. Health Sun
12. HealthLink
13. Amerigroup
14. Medicare
15. Medicaid
16. Or another partner that can provide claims data on participant's behalf

Exclusion Criteria:

-Unable to meet inclusion criteria

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2117 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogel JM, Hung TY, Coughlin E, Delgado F, Kheterpal V, Quer G, Topol E. A Randomized Trial of At-Home COVID-19 Tests, Telemedicine, and Rapid Prescription Delivery for Immunocompromised Individuals. Mayo Clin Proc Innov Qual Outcomes. 2025 May 22;9(3):100627. doi: 10.1016/j.mayocpiqo.2025.100627. eCollection 2025 Jun. PMID 40503088
- See also: Study website — https://immunocare.scripps.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited remotely from across the United States.
Pre-assignment Details: After completing consent, participants verify their eligibility by connecting their health plan or EHR data, or manually sharing information to verify their eligibility. After confirmation of eligibility, participants are randomized into control or intervention arms. Many participants completed enrollment but did not verify their eligibility and therefore are not included in the randomized participants count.
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 495 | 521
Completed | 493 | 517
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: These participants completed the baseline survey where demographics were reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 310 | 285 | 595
Age, Categorical [Count of Participants; unit: Participants] — Participant ages were inferred from their date of birth Population: Ages were reported for all who responded to the baseline survey
  Participants
    number analyzed (Participants) | 292 | 250 | 542
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 88 | 72 | 160
    >=65 years | 204 | 178 | 382
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Nonbinary | 8 | 4 | 12
  Transgender | 0 | 4 | 4
  Prefer not to answer | 0 | 0 | 0
  Woman | 198 | 150 | 348
  Man | 90 | 94 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Middle Eastern | 1 | 0 | 1
  White only | 262 | 218 | 480
  Hispanic only | 5 | 1 | 6
  Black / African American | 3 | 3 | 6
  Other | 1 | 1 | 2
  Multiple races/ethnicities | 12 | 12 | 24
  Prefer not to answer | 3 | 1 | 4
  Asian | 8 | 8 | 16
Primary eligibility category [Count of Participants; unit: Participants] — We analyzed the data based on whether participants primarily met eligibility criteria by being immunocompromised or at least age 65; if a participant was both, they were assigned to the immunocompromised group. Population: This information was collected based on the eligibility verification process and is only presented for participants that shared outcome data. These subgroups are reported on in the analysis.
  Participants
    Immunocompromised | 176 | 160 | 336
    Age 65+ | 134 | 125 | 259

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospitalizations Including COVID Medications
Description: In claims data COVID hospital admissions were defined as: claim type is "HOSP" or "Institutional" or location display contains "inpatient" with COVID diagnosis or COVID procedure or COVID medication in the same medical episode. In survey data, participants were asked to self-report COVID hospitalizations.
Time Frame: During study participation (on average 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 310 | 285
Participants
  COVID medication | 59 | 58
  COVID hospitalization | 15 | 22
  COVID ICU stay | 1 | 13
  No COVID infection reported | 235 | 192

2. Primary Outcome: Cost of Care
Description: Investigators will compare the cost of care for COVID-19 infections between the control and intervention arms.
Time Frame: During study participation (on average 12 months)
Population: Participants with claims and/or survey data were included.
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 310 | 285
dollars | 2,022 [0 to 4,655] | 5,740 [3,107 to 8,373]

ADVERSE EVENTS:
Time Frame: Participants could report an adverse event at any time during their participation.
Description: Participants were able to report adverse events to the study team by email at any time. EHR and claims data were also analyzed for mortality.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/495 | 0/521
Serious Adverse Events (participants affected / at risk) | 0/495 | 0/521
Other Adverse Events (participants affected / at risk) | 0/495 | 0/521

LIMITATIONS AND CAVEATS:
The study ended early because the intervention device's FDA approval was revoked. As a result the study was underpowered and the intervention is no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT05655546/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT05655546/ICF_001.pdf